CLINICAL TRIAL: NCT02545816
Title: A Validation Study to Compare Bispectral Index EEG Monitoring With Full EEG in Patients With an Acute Neurological Insult
Brief Title: Comparing Simplified EEG Monitoring Tool With Standard EEG Monitoring in Patients With Acute Neurological Insult
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, prof. dr. Frank Jans, prof. dr., Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BISZOL1
Record Dates: First submitted 2015-08-20; First posted 2015-09-10 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Acute Neurological Insult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- study group (Other): Patients (age ≥ 18 years) admitted to the ICU with an acute neurological insult which will be sedated/ventilated (Glasgow Coma Scale (GCS) ≤ 8).
  Interventions: Device: Bispectral index (BIS) EEG monitoring

INTERVENTIONS:
Device: Bispectral index (BIS) EEG monitoring — The Bispectral Index (BIS) EEG monitor is a simplified EEG monitoring device which was originally designed to monitor the depth of hypnosis during general anesthesia. It does this by analyzing changes in the processed electroencephalogram (EEG) which occur with the hypnotic state and creating a measure (or index) indicative of these changes. A number between 0 and 100 is derived, with values above 70 associated with an awake state. The monitor also provides a single channel EEG, an electromyogram (EMG) and an index of signal quality (SQI), all in real time.

SUMMARY:
After any acute brain injury, a primary pathophysiological response arises, enabling the brain to develop seizures and/or a status epilepticus (SE). These are frequently reported in patients admitted to the intensive care unit (ICU) with traumatic brain injury and brain injury caused by subarachnoid or intracerebral hemorrhage. Seizures can be presented without any clinical motor signs, which are then termed as nonconvulsive, and therefore remain frequently clinically unrecognized. As such, it is of great importance that these patients are diagnosed as early as possible since the increased metabolic demand and blood flow associated with an epileptic insult may further compromise the brain at risk. Thus far, continuous EEG (cEEG) is the only clinical instrument that is able to detect the development of early epileptic activity. Unfortunately, cEEG is not available in most ICUs and is labor-intensive, expensive and difficult to interpret for non-trained physicians. Therefore, a more simple and prognostic accurate EEG device is highly warranted to detect seizures in an early stage so that patients might benefit from a specific and early treatment. A validation study in comatose patients with an acute neurological insult will be conducted to provide evidence that simplified Bispectral Index EEG monitoring has the potential to detect epileptic activity as reliable as its gold standard, full EEG monitoring. Thereby, BIS EEG monitoring could possibly be used to facilitate the prognostication and management of epileptic seizures in this patient cohort which could eventually improve the clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients (age ≥ 18 years) admitted to the ICU with an acute neurological insult which will be sedated/ventilated (Glasgow Coma Scale (GCS) ≤ 8).
* Ability to place BIS sensors on the forehead
* Written informed consent form has to be obtained from the patient's next of kin and has to be reconfirmed if the patient regains consciousness

Exclusion Criteria:

* Age < 18 years
* Inability to place BIS sensors on the forehead (e.g. due to frontal decompression)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
A comparison between BIS derived EEG and standard full EEG | 15 minutes before or after the acquisition of standard full EEG monitoring.
  Unfiltered BIS derived EEG data from 15 minutes before or after the acquisition of a full intermittent EEG will be used to compare BIS derived EEG traces with full intermittent EEG traces. These data will be (retrospectively) analyzed by experienced neurophysiologists for the presence of seizures and/or status epilepticus.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Jans, prof. dr., Principal Investigator — Ziekenhuis Oost-Limburg, Hasselt University; Cathy De Deyne, prof. dr., Study Chair — Ziekenhuis Oost-Limburg, Hasselt University; Willem Boer, dr., Study Chair — Ziekenhuis Oost-Limburg; Pascal Vanelderen, prof. dr, Study Chair — Ziekenhuis Oost-Limburg, Hasselt University; Ward Eertmans, drs., Study Chair — Hasselt University
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium